CLINICAL TRIAL: NCT03246750
Title: Phase I/II Study of Brentuximab Vedotin and Methotrexate/ L-asparaginase/ Dexamethasone (B-MAD) Chemotherapy in Patients With Newly-diagnosed Extranodal NK/ T-cell Lymphoma
Brief Title: B-MAD Chemotherapy in Newly-diagnosed Extranodal NK/ T-cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Thai Lymphoma Study Group (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Asst.Prof.Udomsak Bunworasate, A.Prof., The Thai Lymphoma Study Group
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLSG-2017-T01
Record Dates: First submitted 2017-07-13; First posted 2017-08-11 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Extranodal NK/T-cell Lymphoma
Keywords: Brentuximab Vedotin
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — Cisplatin

STUDY DESIGN:
Intervention Model Description: 3+3 dose escaltion design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- B-MAD chemotherapy (Experimental): Brentuximab Vedotin, Methotrexate, L-Asparaginase, and Dexamethasone
  Interventions: Drug: B-MAD chemotherapy

INTERVENTIONS:
Drug: B-MAD chemotherapy — B-MAD chemotherapy
  Other Names: Involved field radation, cisplatin

SUMMARY:
Study Title: Phase I/II study of brentuximab vedotin and methotrexate/ L-asparaginase/ dexamethasone (B-MAD) chemotherapy in patients with newly-diagnosed Extranodal NK/T-cell Lymphoma

Phase: I/II

Number of Patients: 36

Study Objectives

Primary

* To determine the safety and optimal dose of brentuximab vedotin when use in combination with methotrexate, L-asparaginase and dexamethasone in the treatment of newly-diagnosed ENKTL patients

Secondary

* To evaluate the clinical efficacy of this regimen
* To access the overall responses including overall response rate (ORR), disease-free survival (DSF), progression-free survival (PFS).

Overview of Study Design:

Open-label, multicenter, non-randomized, 3+3 dose escalation study of brentuximab vedotin in combination with fixed-dose MAD chemotherapy. The first cycle will be evaluated for the determination of the recommended phase II dose.

Patients will be received the treatment according to the stage of disease as follows:

* Patients with localized ENKTL (stage IE or stage IIE) will receive involved-field radiation (IRFT) with concomitant weekly intravenous Cisplatin. Three to five weeks after the completion of IFRT and cisplatin, B-MAD (Brentuximab vedotin, Methotrexate, L-asparaginase and Dexamethasone) regimen will be given every 21 days for 3 cycles.
* Patients with advanced ENKTL (stage III or stag IV) will receive B-MAD every 21 days for 6 cycles.

Study Population:

Patients with newly-diagnosed ENKTL will be screened for enrollment.

Duration of Study: 3 years

DETAILED DESCRIPTION:
Study Title: Phase I/II study of brentuximab vedotin and methotrexate/ L-asparaginase/ dexamethasone (B-MAD) chemotherapy in patients with newly-diagnosed Extranodal NK/T-cell Lymphoma

Phase: I/II

Number of Patients: 36

Study Objectives

Primary

* To determine the safety and optimal dose of brentuximab vedotin when use in combination with methotrexate, L-asparaginase and dexamethasone in the treatment of newly-diagnosed ENKTL patients

Secondary

* To evaluate the clinical efficacy of this regimen
* To access the overall responses including overall response rate (ORR), disease-free survival (DSF), progression-free survival (PFS).

Overview of Study Design:

Open-label, multicenter, non-randomized, 3+3 dose escalation study, starting with 1.2 mg/kg brentuximab vedotin i.v. on day 1 of a 21-day cycle in combination with fixed-dose MAD (Methotrexate, L-asparaginase and Dexamethasone) chemotherapy. The first cycle will be evaluated for the determination of the recommended phase II dose.

Patients will be received the treatment according to the stage of disease as follows:

* Patients with localized ENKTL (stage IE or stage IIE) will receive involved-field radiation (IRFT) 40-50 Gy with concomitant weekly intravenous Cisplatin. Three to five weeks after the completion of IFRT and cisplatin, B-MAD chemotherapy will be given every 21 days for 3 cycles.
* Patients with advanced ENKTL (stage III or stag IV) will receive B-MAD every 21 days for 6 cycles.

Study Population:

Patients with newly-diagnosed ENKTL will be screened for enrollment.

Duration of Study: 3 years

Determination of Sample Size

ENKTL is a rare and highly aggressive disease. Due to the rarity, most published studies evaluating new treatment regimen for ENKTL enrolled approximately 20-40 patients in their studies. Since the phase I of this study is designed as 3+3 dose escalation, then this study will enroll approximately 3-12 patients with localized stage in phase I for dose finding. The beginning dose of brentuximab vedotin will be 1.2 mg/kg, escalating gradually until dose limiting toxicity (DLT) is observed. Initially, 3 patients will be treated with 1.2 mg/kg of brentuximab vedotin and will be monitored for DLT. If there is no DLT observed in all 3 patients at the end of their first treatment cycle, dose escalation to the next dose level (1.8mg/kg) may commence. If there is a DLT observed in 1 of the first 3 patients, additional 3 patients will be included, expanding the cohort to 6 patients. This cohort of patients will be treated with the same previous dose of 1.2 mg/kg and monitor for DLTs. If no DLT observed, dose escalation to the next level (1.8 mg/kg) may commence. If there are DLTs observed in 2 or higher in any of the 6 patients prior dose (0.8mg/kg) will be defined as MTD. There will be no further additional patient inclusion and dose escalation beyond the maximum number of 12 patients and 1.8mg/kg, as MTD will be exceeded.

For phase II study, after reviewed the number of ENKTL patients in the Thai Lymphoma Study Group Registry, there were 106 newly diagnosed ENKTL patients in the registry from 2007-2013. This translated to approximately 15 newly diagnosed ENKTL patients per year. Since this study has the time for patient accruement of three years and with respect to the reference from other previous studies, the total approximate patients in this study for phase I and II is 36.

Populations for Analyses

The full analysis set (FAS) comprises of all patients who were enrolled into the study.

The per-protocol analysis (PAS) set comprises of all patient in the FAS who completed cycles of B-MAD.

The dose-determining set (DDS) comprises of all patients in the SAS who had at least one valid safety assessment after completion of the first cycle of B-MAD or discontinue earlier due to DLT.

Demographic and Baseline Characteristics

Demographic and baseline characteristics will be listed individually by patient, and summarized by cohort using descriptive statistic. The FAS will be used.

Efficacy Analysis

The efficacy analysis set (EAS) comprises of all patients who are able to evaluate for efficacy at least once post-baseline.

Safety Analysis

The safety analysis set (SAS) comprises of all patients of the FAS who received at least one dose of B-MAD and had at least one valid post-baseline safety assessment. (The statement that a patient had no adverse events on the CRF confirms a valid safety assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with previously untreated ENKTL as defined by the World Health Organization (WHO) classification
* Age 18-60 years
* Localized (stage I, II) or advanced (stage III, IV) disease
* Adequate organ function
* Signed informed consent

Exclusion Criteria:

* Patients with other subtypes of non-Hodgkin lymphoma, including myeloid/NK cell precursor acute leukemia, blastic NK cell lymphoma/precursor NK cell lymphoblastic leukemia, aggressive NK cell leukemia, and peripheral T cell lymphoma, unspecified
* Prior chemotherapy or radiotherapy for ENKTL
* Seropositivity for HIV and severe infection
* Prior or other concomitant malignant tumors
* Pregnant or breastfeeding patients
* Evidence of any other disease or medical conditions that contraindicate use of the study drug, or patients at high risk from treatment complications
* Patients suffering from psychiatric disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | At the end of Cycle 1 (each cycle is 21 days)
  Patients will be assessed for dose-limiting toxicity (DLT) during the first cycle.
  DLTs are described as follows:
  For non-hematologic toxicities
  • Any related non-hematologic events of grade 3 or higher, with the exception of:
  * grade 3 fatigue
  * grade 3 or 4 nausea and vomiting lasting than 24 hours
  * grade 3 non-hematologic laboratory abnormalities resolving to grade 1 or baseline within 14 days
  * grade 3 or 4 allergic or hypersensitivity reaction
  For hematologic toxicities
  * Related grade 4 neutropenia lasting > 7 days
  * Related grade 3 febrile neutropenia requiring antibiotics
  * Related grade 4 febrile neutropenia
  * Related grade 4 thrombocytopenia

SECONDARY OUTCOMES:
Treatment responses | At 7th week after last BV dosing
  The treatment response will be evaluated according to the 2014 Recommendations for Initial Evaluation, Staging and Response Assessment of Hodgkin and Non-Hodgkin Lymphoma - The Lugano Classification.
Disease-free survival | 1 year
  Time from complete remission to relapse or death as a result of lymphoma or acute toxicity of treatment
Progression-free survival | 1 year
  Time from entry on to study to disease progression or death as a result of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Udomsak Bunworasate, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No